CLINICAL TRIAL: NCT06195995
Title: Brain Mechanism and Intervention of Executive-control Dysfunction Among Gambling Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JDu-012
Record Dates: First submitted 2023-12-24; First posted 2024-01-08 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2023-12

CONDITIONS: Transcutaneous Electric Nerve Stimulation; Gambling
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group for gambling addiction (Experimental): A 40-minute transcranial alternating current stimulus intervention of real stimulus is conducted twice a day (at least 3 hours apart) for a total of 10 days in the intervention group of gambling addiction.
  Interventions: Device: Transcranial alternating current stimulation-true stimulus

INTERVENTIONS:
Device: Transcranial alternating current stimulation-true stimulus — Three conductive electrodes are placed overhead. In the 10/20 international placement system, a 4.45 9.53 cm electrode is placed on the forehead corresponding to Fpz, Fp1 and Fp2. Two 3.18 3.81 cm electrodes are placed on the mastoid region of each side. The tACS stimulation waveform includes ramp-up and ramp-down periods of 180 and 12 s, respectively. The frequency of stimulation is 77.5Hz, and the current is 15mA.

SUMMARY:
The investigators assume that transcranial Alternating Current Stimulation (tACS) could improve gambling disorder patients' executive-control function by adjusting the synchronization patterns and enhancing the functional connectivity of the prefrontal-ventral striatum pathway. This study intends to test the effect of tACS treatment. Three-month follow-up assessment will be conducted to test the changing of the executive-control function and its mechanism.

DETAILED DESCRIPTION:
Gambling disorder is become a major social and public health problem in China. Executive-control dysfunction is the main symptom of behavioral addiction like gambling disorder. Previous studies have demonstrated the relationship between cognitive dysfunction and prefrontal-ventral striatum pathway. Studies have shown that abnormal phase synchronization and phase-amplitude coupling (PAC) induced the impairment of cognition, and transcranial Alternating Current Stimulation (tACS) could improve executive-control function by adjusting the abnormal synchronization. However, it has not been verified among gambling disorder patients. The investigators assume that tACS could improve gambling disorder patients' executive-control function by adjusting the synchronization patterns and enhancing the functional connectivity of the prefrontal-ventral striatum pathway. This study intends to test the effect of tACS treatment. Three-month follow-up assessment will be conducted to test the changing of the executive-control function and its mechanism. This study will provide a practical and theoretical basis for developing a novel treatment for gambling disorder.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-60, male or female, with 9 or more years of education, and able to complete questionnaire evaluation and behavioral tests
* Meet DSM-5 (Diagnostic and Statistical Manual of mental disorders，DSM) diagnostic criteria for gambling disorder
* Have gambled for at least one year (at least once a week)
* Normal vision and hearing, or within the normal range after correction
* Agree to cooperate in the follow-up evaluation
* No metal implantation in the head, no history of nerve problems or head injury, and no skin sensitivity

Exclusion Criteria:

* Have severe cognitive impairment, such as a history of head trauma, cerebrovascular disease, epilepsy, etc.
* Have used drugs promoting cognitive function in the last 6 months
* Have impaired intelligence (Intelligence Quotient<70)
* Abuse or dependence of psychoactive substances (except nicotine) in the last 5 years

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The change of gambling behavior | baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  Questions including monetary loss, time, frequency and interval of gambling will be answered by patients to quantify their gambling behavior.
The change of gambling craving | baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  Gambling craving will be measured by the gambling craving Visual Analog Scale (VAS). The total score of VAS ranged from 0 to 10, in which higher scores mean a higher level of gambling craving.
The change of gambling symptom | baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  Gambling symptom will be measured by the Gambling Symptom Assessment Scale (G-SAS). The total score of G-SAS ranged from 0 to 48, in which higher scores mean a higher level of gambling symptom.
The change of pathological gambling | baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  Pathological gambling will be measured by the Yale-Brown Obsessive Compulsive Scale adapted for Pathological Gambling (PG-YBOCS). The total score of PG-YBOCS ranged from 0 to 40, in which higher scores mean a higher level of pathological gambling.

SECONDARY OUTCOMES:
The change of self-control | baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  The change of self-control will be measured by the stop-signal task and balloon analog risk-taking task.

OTHER OUTCOMES:
The change of depression | baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  Depression will be measured by the Patient Health Questionnaire-9(PHQ-9). The total score of PHQ-9 ranged from 0 to 27, in which higher scores mean a higher level of depression.
The change of anxiety | baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  Anxiety will be measured by the questionnaire of Generalized Anxiety Disorder(GAD-7). The total score of GAD-7 ranged from 0 to 21, in which higher scores mean a higher level of anxiety.
The change of sleep | baseline, immediately after the intervention, two weeks after the intervention, one month after the intervention, two months after the intervention, three months after the intervention
  Sleep will be measured by the Pittsburgh Sleep Quality Index (PSQI) rated by both patients and observers. The total score of PSQI ranged from 0 to 21, in which higher scores mean a lower level of sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Du, M.D., Ph.D., Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No